CLINICAL TRIAL: NCT00067340
Title: Northwest Alaska Center to Reduce Oral Health Disparity Project 2: Caries Transmission Prevention in Alaska Native Infants
Brief Title: Caries Transmission Prevention in Alaska Native Infants
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit sufficient number of subjects
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, David Grossman, Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19945-C; U54DE014254 (NIH)
Record Dates: First submitted 2003-08-15; First posted 2003-08-20 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2010-04

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Subjects received chlorhexidine mouthwash and xylitol gum , in addition to the usual care specified under the control group
  Interventions: Drug: Chlorhexidine mouth rinse; Other: Xylitol chewing gum
- Control (Placebo Comparator): Subjects received enhanced dental care, health information, toothbrushes and toothpaste. They also received placebo gum and placebo mouth rinse

INTERVENTIONS:
Drug: Chlorhexidine mouth rinse — women received daily chlorhexidine oral rinses for two weeks prior to delivery of the infant.
  Arms: Intervention group
Other: Xylitol chewing gum — Women were asked to chew xylitol chewing gum three times per day following the birth of their infant for up to two years postpartum
  Arms: Intervention group

SUMMARY:
The purpose of this study is to conduct a community based, randomized control trial to determine if the use of chlorhexidine mouth rinse and xylitol-sweetened chewing gum will reduce the vertical transmission of caries between Alaska Native mothers to their infants.

DETAILED DESCRIPTION:
Alaska Native children are disproportionately affected by early childhood caries, compared to all U.S children. Dental care needs for adults and children in rural Alaska far exceed the acute care and prevention resources available. As a result, there is a high level of dental morbidity present among adults that likely contributes to early transmission of mutans streptococci (MS) from adult caregivers to infants in the household. Furthermore, the cultural practice of pre-mastication of solid food for infant feeding amplifies the transmission of oral secretions from adult to child. The prevention of early MS acquisition and subsequent caries in infants and toddlers requires efforts starting at birth. Since Alaska Natives are a rural population at high risk for caries, interruption of vertical transmission of MS using a combination of improved oral hygiene practices, and topical antimicrobials and bacteriostatic agents may be an ideal prevention strategy for childhood caries. Chlorhexidine and xylitol are two agents that have been shown to reduce dental decay and MS counts.

The specific aim of this proposal is to conduct a community based, randomized blinded trial to determine if the serial use of chlorhexidine and xylitol will reduce the vertical transmission of caries between Alaska Native mothers and infants. We hypothesize that a two week period of twice-daily chlorhexidine mouthwash use prior to delivery, followed by a subsequent two year period of maternal xylitol gum use, will lead to a significant reduction in the age-specific prevalence of early childhood caries at 12 and 24 months of age among the offspring of mothers in the intervention group, compared to control group mothers. We also hypothesize that, compared to controls, mothers and children in the intervention group will have significant reductions in oral MS counts at each follow-up interval.

If proven successful, this intervention could have a significant impact on the prevalence of caries among young Alaska Native children and other population groups at high risk for childhood caries.

ELIGIBILITY:
* primiparous or multiparous pregnant Alaska Native mothers of all ages
* in the last month of pregnancy
* reside in the health service delivery area of the native health corporation, in one of the communities with the highest birth counts from 2002
* eligible for obstetric care from the health corporation
* plan to give birth to their infant in a specified city of Alaska

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2003-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Grossman, MD MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States